CLINICAL TRIAL: NCT07125404
Title: Effectiveness of Low-Level Laser Auriculotherapy in the Treatment of Myogenic Temporomandibular Disorders and Anxiety: A Randomized Clinical Trial
Brief Title: Low-Level Laser Auriculotherapy in the Treatment of Myogenic Temporomandibular Disorders and Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quiropraxia y Equilibrio (Other)
Responsible Party: Principal Investigator, Hernán Andrés de la Barra Ortiz, PhD., Quiropraxia y Equilibrio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06082025
Record Dates: First submitted 2025-08-06; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Temporomandibular Disorder; Anxiety State
Keywords: Laser Therapy; Low-level Light Therapy; Auriculotherapy; Joint Disorders; Temporomandibular Joint Dysfunction Syndrome; Anxiety
MeSH Terms: conditions — Temporomandibular Joint Disorders; Anxiety Disorders; Joint Diseases; Temporomandibular Joint Dysfunction Syndrome | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Parallel-group, randomized, placebo-controlled trial with participant and assessor blinding
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLLT-AT (Experimental): Participants will receive low-level laser auriculotherapy (LLLT-AT) using an infrared class IIIb diode laser (905 nm). The laser will be applied to four auricular acupuncture points: Shenmen (TF4), Kidney (AH9), Liver (AH11), and Point Zero (O'), following the protocol by Marques et al. (2023). Each point will receive 4 J of energy (total of 16 J per session) with an average output power of 71 mW over 224 seconds. The treatment will be applied to the auricle ipsilateral to the symptomatic TMJ or to the more painful side in bilateral cases. In addition to LLLT-AT, the experimental group will receive a baseline manual therapy treatment consisting of bilateral myofascial release of the masseter and temporalis muscles. A total of six sessions will be delivered over a period of three weeks.
  Interventions: Radiation: Low-level laser auriculotherapy (LLLT-AT); Other: Myofascial release
- Sham LLLT-AT (Sham Comparator): Participants in the sham laser group will be treated under the same conditions as the experimental group, using the same device (COMBI 400L, Gymna®), dosage parameters, and safety procedures. However, a simulated laser emission will be used by disconnecting the probe, thereby preventing the laser beam from being emitted. The laser will be applied to the same four auricular points as in the experimental group. This sham condition is unlikely to be perceived by participants, as low-level laser therapy is athermal and does not produce noticeable sensations during application. In addition to sham LLLT-AT, this group will receive a baseline manual therapy treatment consisting of bilateral myofascial release of the masseter and temporalis muscles. A total of six sessions will be delivered over a period of three weeks.
  Interventions: Other: Sham Low-level laser auriculotherapy (sham LLLT-AT); Other: Myofascial release

INTERVENTIONS:
Radiation: Low-level laser auriculotherapy (LLLT-AT) — Low-Level Laser Auriculotherapy (LLLT-AT) is a non-invasive, painless treatment that applies infrared laser (class IIIb, 905 nm) to specific auricular acupuncture points. It aims to reduce musculoskeletal pain and anxiety by stimulating mitochondrial cytochrome c oxidase, increasing ATP production, promoting tissue repair, and modulating inflammation. LLLT also reduces nerve excitability and triggers β-endorphin release, aiding in pain control. Auricular stimulation may influence autonomic nervous system activity, impacting both physical and emotional symptoms. The intervention consists of two sessions per week over three weeks, following standard laser safety procedures.
  Other Names: Laser Auriculotherapy; Auricular Photobiomodulation Therapy
  Arms: LLLT-AT
Other: Sham Low-level laser auriculotherapy (sham LLLT-AT) — Sham LLLT-AT replicates the active procedure using the same laser device and parameters, but without light emission. The probe will be deactivated and applied to the same auricular points twice weekly for three weeks. As LLLT is painless and athermal, participants are unlikely to distinguish the sham condition. Standard safety protocols will be maintained.
  Other Names: Sham Laser auriculotherapy; Sham Auricular Photobiomodulation Therapy
  Arms: Sham LLLT-AT
Other: Myofascial release — Myofascial release is a manual therapy applied bilaterally to the masseter and temporalis muscles as a baseline intervention. Each session includes 1 minute of ischemic pressure, 1 minute of myofascial release, 30 seconds of positional release, and 30 seconds of general mobilization per muscle. The protocol consists of two sessions per week for three weeks (six sessions total), aiming to reduce muscle tension and improve mandibular function.

SUMMARY:
Summary:

Low-level laser auriculotherapy (LLLT-AT) is a non-invasive technique that has gained attention for managing musculoskeletal pain and anxiety. Given the painful and emotional components of temporomandibular disorders (TMD), LLLT-AT may offer therapeutic benefits by stimulating auricular points associated with pain modulation and anxiety reduction. This randomized, placebo-controlled, two-arm clinical trial with blinded outcome assessors aims to evaluate the effects of LLLT-AT in individuals diagnosed with myogenic TMD (Axis I, Group I of the DC/TMD classification) and anxiety. The study will be conducted at the Physical Agents Laboratory of Universidad Andrés Bello. Eligible participants will include members of the university community with myogenic TMD (Axis I, Group I of the DC/TMD classification) and anxiety. Participants will be stratified by sex and randomly assigned to either an experimental group receiving LLLT-AT combined with a standardized myofascial release protocol or a control group receiving sham LLLT-AT with the same myofascial protocol. Interventions will be administered twice weekly for three weeks. Outcome measures will be collected at baseline, post-intervention, and at a four-week follow-up. Primary outcomes include pressure pain threshold (PPT), assessed by algometry, and anxiety level, measured using the GAD-7 scale. Secondary outcomes include maximum mouth opening range of motion (MMOROM) and mandibular functional limitation (MFL), assessed using the Jaw Functional Limitation Scale 8 (JFLS-8).

DETAILED DESCRIPTION:
Material and Methods

1. Study design:

   A double-blind, randomized, placebo-controlled trial with two parallel groups.
2. Study population:

   Participants will include students, faculty, and administrative staff from Universidad Andrés Bello, Casona de Las Condes Campus. Recruitment will be conducted through institutional channels such as bulletin boards, digital posters, and official emails. Interested individuals will be invited for an in-person screening at the Physical Agents Laboratory (KIN 401, Building C5) of the School of Rehabilitation Sciences. The screening will involve a study explanation, eligibility assessment, and a physical examination conducted by an experienced physiotherapist to confirm a myogenic temporomandibular disorder (Axis I, Group I, DC/TMD classification).
3. Sample size and randomization:

   Sample size will be calculated using G*Power® software, assuming a statistical power of 80% (1-β), a significance level of 0.05 (α), a 95% confidence level, and an estimated effect size of 1.0. This value is based on the study by Sancakli et al. (see reference), who reported an increase in the pressure pain threshold (PPT) of the masseter muscle in patients with myogenic temporomandibular disorders following four weeks of treatment with low-level laser therapy (LLLT). The minimum estimated sample size is 28 participants, 14 per group (LLLT-AT plus myofascial release and sham LLLT-AT plus myofascial release). To account for potential data loss or participant dropout during the study, researchers will apply a 15% increase to the calculated sample size. This decision aligns with item 8 of the Physiotherapy Evidence Database (PEDro) scale, which requires that outcome measures be obtained from at least 85% of participants. Therefore, a minimum of 16 participants per group will be recruited.

   Selected participants will be allocated into two groups through a simple randomization process: experimental group (LLLT-AT) and control group (sham LLLT-AT). Additionally, stratification by sex will be performed to ensure an equal proportion of male and female participants in each group. Randomization will be carried out using the web-based tool Research Randomizer (https://www.randomizer.org/). FFollowing the laser intervention, both the experimental and control groups will receive bilateral myofascial release treatment targeting the masticatory muscles (masseter and temporalis) (35). Participants will be blinded to group allocation.
4. Selection criteria

   * Inclusion Criteria: Participants must be ≥18 years old, of any gender, with a clinical diagnosis of unilateral or bilateral myogenic temporomandibular disorder (TMD) based on DC/TMD criteria. This includes spontaneous or palpation-induced myalgia in the masticatory muscles. Participants must have experienced at least one episode of local, referred, or radiating masticatory pain in the past 30 days lasting at least one hour. A GAD-7 score of ≥5 is also required.
   * Exclusion Criteria: Recent musculoskeletal injuries in the cervical region; skin lesions or diseases on the auricle; regular use of medications such as corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs), or photosensitizing agents (e.g., tetracyclines, quinolones, or sulfonamides); tattoos on or near the auricular region; history of cancer or tumors within the past five years; Fitzpatrick skin phototypes V-VI; autoimmune diseases (e.g., lupus erythematosus, hepatic porphyria, or pellagra); and epilepsy.
   * Discontinuation Criteria: Participants who fail to complete the evaluation or treatment protocol due to withdrawal or non-attendance will be excluded from the final analysis.
5. Interventions:

   The experimental group will receive two weekly sessions of low-level laser auriculotherapy (LLLT-AT), while the control group will receive two weekly sessions of sham LLLT-AT. Sessions will be scheduled with a two-day interval between each session. Both groups will receive a standard manual therapy protocol consisting of bilateral myofascial release of the masseter and temporalis muscles. A total of six treatment sessions will be administered over three weeks.
   * LLLT-AT Procedure. The experimental group will be treated with low-level laser auriculotherapy using an infrared low-power diode laser (class IIIb) with a wavelength of 905 nm. LLLT-AT will be applied to four auricular acupuncture points: Shenmen (TF4), Kidney (AH9), Liver (AH11), and Point Zero (O'). The protocol proposed by Marques et al. (2023) will be followed, delivering 4 joules (J) of energy per point. Treatment parameters include a mean output power of 71 milliwatts (mW) and an irradiation time of 56 seconds per point (total application time: 224 seconds), resulting in a total energy dose of 16 J per session. LLLT-AT will be applied to the auricle ipsilateral to the symptomatic temporomandibular joint (TMJ). In cases of bilateral pain, the side with the greater self-reported pain will be treated. Sessions will be performed with the participant in the lateral decubitus position, exposing the treated ear. Both the participant and the therapist will wear protective laser goggles during the procedure. The laser device used will be the Combi 400L by GYMNA®.
   * Sham LLLT-AT. In the sham laser group, participants will be treated under the same conditions as the experimental group, using the same equipment (Gymna® COMBI 400L laser), identical dosing parameters, and the same procedural precautions. However, a simulated laser emission will be applied by disconnecting the laser probe, thus preventing beam delivery. This condition will be difficult for participants to detect, as LLLT is an athermal intervention and does not produce perceptible sensations during application.
   * Myofascial Release. Both groups will receive a standard manual therapy intervention based on bilateral myofascial release techniques applied to the masticatory muscles (masseter and temporalis) following this protocol: (A) Temporalis muscle relaxation: Ischemic compression of the trigger point (1 minute), myofascial release of the trigger point (1 minute), positional release (30 seconds), and global myofascial release of the temporalis muscle (30 seconds); (B) Masseter muscle relaxation: Ischemic compression of the trigger point (1 minute), myofascial release of the trigger point (1 minute), positional release (30 seconds), and global myofascial release of the masseter muscle (30 seconds).
6. Outcome Measures:

   Primary outcomes will include changes in pressure pain threshold (PPT) and anxiety level (AL). Secondary outcomes will include changes in maximum mandibular opening range of motion (MMOROM) and mandibular functional limitation (MFL). All assessments will be performed by a blinded independent evaluator. PPT will be measured using algometry at two bilateral points associated with the masseter and temporalis muscles. AL, MMOROM, and MFL will be assessed using the Generalized Anxiety Disorder 7-item scale (GAD-7), a millimeter ruler, and the 8-item Jaw Functional Limitation Scale (JFLS-8), respectively. Assessments will be conducted at three time points: baseline (T0), post-treatment (T1: after the 6th LLLT-AT session, end of week 3), and follow-up (T2: 4 weeks after the end of treatment).
   * PPT. PPT will be measured using a WAGNER FPX® pressure algometer. Assessments will be performed with the participant in a supine position. Four bilateral muscle sites (masseter and temporalis) will be evaluated. Each site will be measured three times with 30-second intervals; the average will be calculated per site. The total PPT will be the sum of the four site averages, expressed in lb/cm². To assess intra-rater reliability, the intraclass correlation coefficient (ICC) will be calculated using repeated PPT measurements at the upper trapezius midpoint in 13 healthy volunteers, with a 48-hour interval.
   * AL. Anxiety will be assessed using the GAD-7 scale, a 7-item Likert questionnaire scored 0-3 per item (Appendix 5). The total score (range: 0-21) reflects anxiety severity. The GAD-7 has been validated in Spanish, with sensitivity = 0.83 and specificity = 0.46 (30,43).
   * MMOROM.The measurement was conducted in the supine position using a millimeter ruler. Researchers will record the distance between the upper and lower central incisors at maximum mouth opening.
   * MFL. The Jaw Functional Limitation Scale (JFLS-8), an 8-item Likert scale (0-10 per item) covering chewing, mouth opening, and communication tasks, will be used to assess the MFL. The maximum score will be used. The JFLS-8 is validated in Spanish and has high reliability (ICC = 0.94-0.96) with a strong correlation to the 20-item version (r = 0.86).
7. Variables

   Conceptual Definition of Study Variables:
   * PPT. The amount of pressure applied to the bellies of the masticatory muscles (masseter and temporalis) that the participant perceives as painful.
   * AL. The degree of tension and/or worry reported by the participant in the past two weeks, framed within the definition of generalized anxiety disorder.
   * MMOROM. The extent or range of movement demonstrated by the participant during maximal mouth opening.
   * MFL. The restriction in the ability of the jaw to perform daily activities such as speaking, smiling, eating, or other functions.
   * LLLT-AT. A therapeutic intervention involves applying laser light with a power below 0.5 watts (W) to specific points on the auricle, which are associated with pain and anxiety modulation.
   * Myofascial Release: A bilateral manual therapy intervention applied to the masticatory muscles (masseter and temporalis).

   Operational Definition of Study Variables:
   * PPT. The PPT will be measured using pressure algometry with a WAGNER FPX algometer. PPT values will be recorded in pounds per square centimeter (lb/cm²).
   * AL. The GAD-7 will be used for assessment. This Likert-scale instrument consists of 7 items scored from 0 to 3. Higher scores indicate greater anxiety severity. The total score classifies anxiety into four categories: no anxiety (0-4), mild (5-9), moderate (10-14), and severe (15-21).
   * MMOROM. The measurement will be done in millimeters using a 10-cm ruler. The evaluator will record the distance between the incisal edges of the upper and lower central incisors during maximal mouth opening.
   * MFL. The JFLS-8 is used to measure MFL. Each item is rated on a 0-10 Likert scale; higher scores indicate greater functional limitation.
   * LLLT-AT. The treatment will be administered using an infrared laser with a wavelength of 905 nm and a power output of 71 mW, which delivers 4 joules (J) of energy per point. The device used will be the Combi 400L (GYMNA®).
   * Myofascial Release: A bilateral treatment will be applied to the masseter and temporalis muscles, consisting of the following sequence: trigger point pressure (1 min), trigger point myofascial release (1 min), positional release (30 sec), and general muscle myofascial release (30 sec).

   Study Variable Type
   * PPT. Dependent variable; continuous quantitative.
   * AL. Dependent variable; ordinal qualitative.
   * MMOROM. Dependent variable; continuous quantitative.
   * MFL. Dependent variable; ordinal qualitative.
   * LLLT-AT. Independent variable; continuous quantitative.
   * Myofascial Release: Independent variable; nominal qualitative.
8. Study phases

   The study will be conducted in three phases:

   - Phase 1 - Screening (2 weeks): A digital screening questionnaire will be distributed to the target population to identify potentially eligible participants. Responses will be reviewed to assess initial eligibility based on inclusion criteria. Individuals who meet the criteria will be contacted and invited to participate. Written informed consent will be obtained prior to enrollment.

   - Phase 2 - Baseline Assessment (2 weeks): Participants will undergo a standardized physical examination to confirm the presence of myogenic TMD, based on the DC/TMD diagnostic criteria. A trained physiotherapist will perform bilateral palpation of the masseter and temporalis muscles. Those presenting localized or referred pain during palpation will be considered eligible. Participants with positive findings will complete the GAD-7 questionnaire to assess anxiety levels.

   - Phase 3 - Intervention and Follow-up (3 weeks + 4-week follow-up): Eligible participants will be randomly assigned to one of two groups: (1) an experimental group receiving LLLT-AT and (2) a control group receiving sham LLLT-AT. Both groups will also receive standardized bilateral myofascial release of the masseter and temporalis muscles. Treatment will be delivered twice per week for three weeks. Primary and secondary outcomes-including PPT, AL, MMOROM, and MFL-will be assessed at baseline, after the intervention, and at 4-week follow-up. All evaluations will be conducted by a blinded assessor, and data will be recorded and managed using Microsoft Excel®.
9. Statistical Analysis Descriptive statistics will be presented for demographic and outcome variables-PPT, AL, MMOROM, and MFL-using measures of central tendency and dispersion: means with standard deviations (mean ± SD) or medians with interquartile ranges (median, IQR), depending on data distribution. Normality will be assessed using the Shapiro-Wilk test. A summary table of participant demographic characteristics will be created and stratified by group. For secondary variables such as sex and body mass index, frequencies and either means or medians will be reported, as appropriate.

For inferential analysis, parametric or non-parametric tests will be selected based on the normality assessment. If normal distribution is confirmed, a two-way ANOVA (factors: group and time) will be applied. If data are non-normally distributed, the Kruskal-Wallis test will be used. Post-hoc analyses will be conducted using Bonferroni or Tukey corrections, as appropriate to the primary test used.

All analyses will be performed using IBM SPSS Statistics version 26, with the significance level set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Clinical diagnosis of unilateral or bilateral myogenic temporomandibular disorder (TMD) based on DC/TMD criteria.
* Presence of myalgia or myofascial pain in the masticatory muscles, either spontaneous or induced by clinical palpation.
* At least one episode of local, referred, or radiating masticatory pain in the past 30 days, lasting at least one hour.
* Score ≥ 5 on the Generalized Anxiety Disorder 7-item scale (GAD-7), indicating generalized anxiety.

Exclusion Criteria:

* Recent musculoskeletal injury in the cervical region.
* Skin lesions or dermatological conditions on the auricle.
* Regular use of medications such as corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs), or photosensitizing agents (e.g., tetracyclines, quinolones, sulfonamides).
* Tattoos on or near the auricular area.
* History of cancer or tumors within the past five years.
* Fitzpatrick skin phototype V or VI.
* Autoimmune diseases (e.g., lupus erythematosus, hepatic porphyria, pellagra).
* Epilepsy.

Discontinuation Criteria

- The participant's withdrawal or non-attendance results in the failure to complete the evaluation or treatment protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain pressure thereshold (PPT) | Baseline, 3 weeks (6 sessions) and 4 weeks (follow-up)
  PPT will be assessed via algometry with the participant in a supine position. Four bilateral points on the masseter and temporalis muscles will be evaluated. Each point will be measured three times with 30-second intervals, and the average of each set will be calculated. The final PPT score will be the sum of the four-point averages, expressed in lb/cm². Data will be recorded in Microsoft Excel®.
Anxiety level (AL) | Baseline, 3 weeks (6 sessions) and 4 weeks (follow-up)
  AL will be assessed using the GAD-7 scale, a validated 7-item questionnaire scored from 0 to 3. It measures anxiety symptoms over the past month, with higher total scores indicating greater severity. The total score (0-21) will be calculated by summing all item responses. The GAD-7 is validated in Spanish and has demonstrated good sensitivity (0.83) and moderate specificity (0.46).

SECONDARY OUTCOMES:
Maximum mandibular opening range of motion (MMOROM) | Baseline, 3 weeks (6 sessions) and 4 weeks (follow-up)
  MMOROM will be measured with the participant in a supine position, head in neutral alignment. The distance between the incisal edges of the upper and lower central incisors during maximum mouth opening will be recorded using a millimeter ruler.
Mandibular functional limitation (MFL) | Baseline, 3 weeks (6 sessions) and 4 weeks (follow-up)
  MFL will be assessed using the JFLS-8, an 8-item Likert-scale questionnaire measuring limitations in jaw function, including chewing, mouth opening, and verbal/non-verbal communication. Each item is scored from 0 (no limitation) to 10 (severe limitation). The total score will reflect the maximum reported limitation. The scale is validated in Spanish and has high reliability (ICC = 0.94-0.96) and strong correlation with the 20-item version (r = 0.86).

CONTACTS AND LOCATIONS:
Overall Officials: Hernán A de la Barra, PhD., Principal Investigator — Exercise and Rehabilitation Sciences Institute, School of Physical Therapy, Faculty of Rehabilitation Sciences, Universidad Andres Bello, Santiago 7591538, Chile
Locations (1):
- Universidad Andrés Bello, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] List T, Jensen RH. Temporomandibular disorders: Old ideas and new concepts. Cephalalgia. 2017 Jun;37(7):692-704. doi: 10.1177/0333102416686302. Epub 2017 Jan 9. PMID 28068790
- [Background] Palmer J, Durham J. Temporomandibular disorders. BJA Educ. 2021 Feb;21(2):44-50. doi: 10.1016/j.bjae.2020.11.001. Epub 2020 Dec 24. No abstract available. PMID 33889429
- [Background] Zielinski G, Pajak-Zielinska B, Ginszt M. A Meta-Analysis of the Global Prevalence of Temporomandibular Disorders. J Clin Med. 2024 Feb 28;13(5):1365. doi: 10.3390/jcm13051365. PMID 38592227
- [Background] Alrizqi AH, Aleissa BM. Prevalence of Temporomandibular Disorders Between 2015-2021: A Literature Review. Cureus. 2023 Apr 2;15(4):e37028. doi: 10.7759/cureus.37028. eCollection 2023 Apr. PMID 37143640
- [Background] Yap AU, Lai YC, Ho HCW. Prevalence of temporomandibular disorders and their associated factors in Confucian heritage cultures: A systematic review and meta-analysis. J Oral Rehabil. 2024 Oct;51(10):2169-2194. doi: 10.1111/joor.13779. Epub 2024 Jun 14. PMID 38873743
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Dos Santos EA, Peinado BRR, Frazao DR, Ne YGS, Fagundes NCF, Magno MB, Maia LC, Lima RR, de Souza-Rodrigues RD. Association between temporomandibular disorders and anxiety: A systematic review. Front Psychiatry. 2022 Oct 13;13:990430. doi: 10.3389/fpsyt.2022.990430. eCollection 2022. PMID 36311527
- [Background] Paludo B, Trevizan PC, Boamah NAA, Rigo L. Prevalence of Temporomandibular Disorder and its association with anxiety in academics: a cross-sectional study. Sao Paulo Med J. 2024 Dec 20;143(1):e2023338. doi: 10.1590/1516-3180.2023.0338.R2.03072024. eCollection 2024. PMID 39774730
- [Background] Lagana G, Malara A, Koumoulis A, Tepedino M, Venza N, Cozza P. Bruxism, perceived anxiety and stress in university students. J Biol Regul Homeost Agents. 2021 Mar-Apr;35(2):787-790. doi: 10.23812/20-578-L. No abstract available. PMID 33934593
- [Background] West KL, Huzij T. A systematic review of manual therapy modalities and anxiety. J Osteopath Med. 2024 Jun 24;124(11):487-497. doi: 10.1515/jom-2024-0001. eCollection 2024 Nov 1. PMID 38905700
- [Background] Ouanounou A, Goldberg M, Haas DA. Pharmacotherapy in Temporomandibular Disorders: A Review. J Can Dent Assoc. 2017 Jul;83:h7. PMID 29513209
- [Background] Fernandez-de-Las-Penas C, Von Piekartz H. Clinical Reasoning for the Examination and Physical Therapy Treatment of Temporomandibular Disorders (TMD): A Narrative Literature Review. J Clin Med. 2020 Nov 17;9(11):3686. doi: 10.3390/jcm9113686. PMID 33212937
- [Background] Craciun MD, Geman O, Leuciuc FV, Holubiac IS, Gheorghita D, Filip F. Effectiveness of Physiotherapy in the Treatment of Temporomandibular Joint Dysfunction and the Relationship with Cervical Spine. Biomedicines. 2022 Nov 17;10(11):2962. doi: 10.3390/biomedicines10112962. PMID 36428529
- [Background] Gauer RL, Semidey MJ. Diagnosis and treatment of temporomandibular disorders. Am Fam Physician. 2015 Mar 15;91(6):378-86. PMID 25822556
- [Background] Vieira A, Reis AM, Matos LC, Machado J, Moreira A. Does auriculotherapy have therapeutic effectiveness? An overview of systematic reviews. Complement Ther Clin Pract. 2018 Nov;33:61-70. doi: 10.1016/j.ctcp.2018.08.005. Epub 2018 Aug 23. PMID 30396628
- [Background] Vieira A, Sousa P, Moura A, Lopes L, Silva C, Robinson N, Machado J, Moreira A. The Effect of Auriculotherapy on Situational Anxiety Trigged by Examinations: A Randomized Pilot Trial. Healthcare (Basel). 2022 Sep 21;10(10):1816. doi: 10.3390/healthcare10101816. PMID 36292262
- [Background] Choi SY, Kim YJ, Kim B. [Effect of Auriculotherapy on Musculoskeletal Pain: A Systematic Review and Meta-Analysis]. J Korean Acad Nurs. 2022 Feb;52(1):4-23. doi: 10.4040/jkan.21121. Korean. PMID 35274617
- [Background] Lee EJ. Effects of auriculotherapy on addiction: a systematic review. J Addict Dis. 2022 Jul-Sep;40(3):415-427. doi: 10.1080/10550887.2021.2016011. Epub 2022 Feb 18. PMID 35179436
- [Background] Clijsen R, Brunner A, Barbero M, Clarys P, Taeymans J. Effects of low-level laser therapy on pain in patients with musculoskeletal disorders: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2017 Aug;53(4):603-610. doi: 10.23736/S1973-9087.17.04432-X. Epub 2017 Jan 30. PMID 28145397
- [Background] de la Barra Ortiz HA, Arias M, Meyer von Schauensee M, Liebano RE. Efficacy of High-intensity laser therapy in patients with temporomandibular joint disorders: A systematic review and meta-analysis. Lasers Med Sci. 2024 Aug 7;39(1):210. doi: 10.1007/s10103-024-04162-4. PMID 39112804
- [Background] Cotler HB, Chow RT, Hamblin MR, Carroll J. The Use of Low Level Laser Therapy (LLLT) For Musculoskeletal Pain. MOJ Orthop Rheumatol. 2015;2(5):00068. doi: 10.15406/mojor.2015.02.00068. Epub 2015 Jun 9. PMID 26858986
- [Background] Marques SL, Ramos AC da S, Boggiss ÉA, de Lima RA, Pinheiro-Araújo CF, Santos ATS, et al. The effect of photobiomodulation auriculotherapy in the treatment of temporomandibular disorders: A double-blind randomized feasibility study. J Photochem Photobiol. 2023 Dec 1;18:100210.
- [Background] Sampaio-Filho H, Bussadori SK, Goncalves MLL, da Silva DFT, Borsatto MC, Tortamano IP, Longo PL, Pavani C, Fernandes KPS, Mesquita-Ferrari RA, Horliana ACRT. Low-level laser treatment applied at auriculotherapy points to reduce postoperative pain in third molar surgery: A randomized, controlled, single-blinded study. PLoS One. 2018 Jun 19;13(6):e0197989. doi: 10.1371/journal.pone.0197989. eCollection 2018. PMID 29920521
- [Background] Menezes FDS, Chaves ECL, Mantuani APA, Marino LS, Alcantara MAR, Nassif MS, de Castro Moura C, Carvalho LC, Iunes DH. Effects of low-power laser auriculotherapy on chronic spinal pain: Randomized clinical trial. Complement Ther Clin Pract. 2022 Aug;48:101578. doi: 10.1016/j.ctcp.2022.101578. Epub 2022 Mar 29. PMID 35405631
- [Background] Butcher NJ, Monsour A, Mew EJ, Chan AW, Moher D, Mayo-Wilson E, Terwee CB, Chee-A-Tow A, Baba A, Gavin F, Grimshaw JM, Kelly LE, Saeed L, Thabane L, Askie L, Smith M, Farid-Kapadia M, Williamson PR, Szatmari P, Tugwell P, Golub RM, Monga S, Vohra S, Marlin S, Ungar WJ, Offringa M. Guidelines for Reporting Outcomes in Trial Reports: The CONSORT-Outcomes 2022 Extension. JAMA. 2022 Dec 13;328(22):2252-2264. doi: 10.1001/jama.2022.21022. PMID 36511921
- [Background] Chan AW, Boutron I, Hopewell S, Moher D, Schulz KF, Collins GS, Tunn R, Aggarwal R, Berkwits M, Berlin JA, Bhandari N, Butcher NJ, Campbell MK, Chidebe RCW, Elbourne DR, Farmer AJ, Fergusson DA, Golub RM, Goodman SN, Hoffmann TC, Ioannidis JPA, Kahan BC, Knowles RL, Lamb SE, Lewis S, Loder E, Offringa M, Ravaud P, Richards DP, Rockhold FW, Schriger DL, Siegfried NL, Staniszewska S, Taylor RS, Thabane L, Torgerson DJ, Vohra S, White IR, Hrobjartsson A. SPIRIT 2025 statement: Updated guideline for protocols of randomised trials. PLoS Med. 2025 Apr 28;22(4):e1004589. doi: 10.1371/journal.pmed.1004589. eCollection 2025 Apr. PMID 40294521
- [Background] Shrestha B, Dunn L. The Declaration of Helsinki on Medical Research involving Human Subjects: A Review of Seventh Revision. J Nepal Health Res Counc. 2020 Jan 21;17(4):548-552. doi: 10.33314/jnhrc.v17i4.1042. PMID 32001865
- [Background] Bhaskar SB. Clinical trial registration: A practical perspective. Indian J Anaesth. 2018 Jan;62(1):10-15. doi: 10.4103/ija.IJA_761_17. PMID 29416145
- [Background] Leskinen J, Suvinen T, Teerijoki-Oksa T, Kemppainen P, Napankangas R, Alstergren P, Le Bell Y, Forssell H, Myllykangas R, Tolvanen M, Doepel M, Sipila K. Diagnostic criteria for temporomandibular disorders (DC/TMD): interexaminer reliability of the Finnish version of Axis I clinical diagnoses. J Oral Rehabil. 2017 Jul;44(7):493-499. doi: 10.1111/joor.12516. Epub 2017 May 6. PMID 28407454
- [Background] Johnson SU, Ulvenes PG, Oktedalen T, Hoffart A. Psychometric Properties of the General Anxiety Disorder 7-Item (GAD-7) Scale in a Heterogeneous Psychiatric Sample. Front Psychol. 2019 Aug 6;10:1713. doi: 10.3389/fpsyg.2019.01713. eCollection 2019. PMID 31447721
- [Background] Coleman W, Mariwalla K, Grimes P. Updating the Fitzpatrick Classification: The Skin Color and Ethnicity Scale. Dermatol Surg. 2023 Aug 1;49(8):725-731. doi: 10.1097/DSS.0000000000003860. Epub 2023 Jul 4. PMID 37523593
- [Background] Kang H. Sample size determination and power analysis using the G*Power software. J Educ Eval Health Prof. 2021;18:17. doi: 10.3352/jeehp.2021.18.17. Epub 2021 Jul 30. PMID 34325496
- [Background] Sancakli E, Gokcen-Rohlig B, Balik A, Ongul D, Kipirdi S, Keskin H. Early results of low-level laser application for masticatory muscle pain: a double-blind randomized clinical study. BMC Oral Health. 2015 Oct 23;15(1):131. doi: 10.1186/s12903-015-0116-5. PMID 26496720
- [Background] Cashin AG, McAuley JH. Clinimetrics: Physiotherapy Evidence Database (PEDro) Scale. J Physiother. 2020 Jan;66(1):59. doi: 10.1016/j.jphys.2019.08.005. Epub 2019 Sep 11. No abstract available. PMID 31521549
- [Background] Lim CY, In J. Randomization in clinical studies. Korean J Anesthesiol. 2019 Jun;72(3):221-232. doi: 10.4097/kja.19049. Epub 2019 Apr 1. PMID 30929415
- [Background] Urbanski P, Trybulec B, Pihut M. The Application of Manual Techniques in Masticatory Muscles Relaxation as Adjunctive Therapy in the Treatment of Temporomandibular Joint Disorders. Int J Environ Res Public Health. 2021 Dec 8;18(24):12970. doi: 10.3390/ijerph182412970. PMID 34948580
- [Background] Wirz-Ridolfi A. The History of Ear Acupuncture and Ear Cartography: Why Precise Mapping of Auricular Points Is Important. Med Acupunct. 2019 Jun 1;31(3):145-156. doi: 10.1089/acu.2019.1349. Epub 2019 Jun 17. PMID 31297168
- [Background] Fisch G, Finke A, Ragonese J, Dugas L, Wrzosek M. Outcomes of physical therapy in patients with temporomandibular disorder: a retrospective review. Br J Oral Maxillofac Surg. 2021 Feb;59(2):145-150. doi: 10.1016/j.bjoms.2020.08.068. Epub 2020 Aug 20. PMID 33280944
- [Background] Aguiar ADS, Nogueira Carrer HC, de Lira MR, Martins Silva GZ, Chaves TC. Patient-Reported Outcome Measurements in Temporomandibular Disorders and Headaches: Summary of Measurement Properties and Applicability. J Clin Med. 2021 Aug 26;10(17):3823. doi: 10.3390/jcm10173823. PMID 34501273
- [Background] Ohrbach R, Larsson P, List T. The jaw functional limitation scale: development, reliability, and validity of 8-item and 20-item versions. J Orofac Pain. 2008 Summer;22(3):219-30. PMID 18780535
- [Background] Sanches ML, Juliano Y, Novo NF, Guimaraes AS, Rodrigues Conti PC, Alonso LG. Correlation between pressure pain threshold and pain intensity in patients with temporomandibular disorders who are compliant or non-compliant with conservative treatment. Oral Surg Oral Med Oral Pathol Oral Radiol. 2015 Oct;120(4):459-68. doi: 10.1016/j.oooo.2015.05.017. Epub 2015 May 29. PMID 26188733
- [Background] Rampazo da Silva EP, Silva VR, Bernardes AS, Matuzawa F, Liebano RE. Segmental and extrasegmental hypoalgesic effects of low-frequency pulsed current and modulated kilohertz-frequency currents in healthy subjects: randomized clinical trial. Physiother Theory Pract. 2021 Aug;37(8):916-925. doi: 10.1080/09593985.2019.1650857. Epub 2019 Aug 12. PMID 31402740
- [Background] Vrublevska J, Renemane L, Kivite-Urtane A, Rancans E. Validation of the generalized anxiety disorder scales (GAD-7 and GAD-2) in primary care settings in Latvia. Front Psychiatry. 2022 Oct 6;13:972628. doi: 10.3389/fpsyt.2022.972628. eCollection 2022. PMID 36276320
- [Background] Sun R, Liu T, Liu Y, Zhang S, Yue Y, Jiang N, Zhang L, Xiong X. Simplified Jaw Functional Limitation Scale for Temporomandibular Disorders: Psychometric Evaluation. Oral Dis. 2025 Jun;31(6):1854-1860. doi: 10.1111/odi.15253. Epub 2025 Jan 10. PMID 39791447